CLINICAL TRIAL: NCT05046626
Title: Effect of Intervention Based on Nutritional Counseling on Changes in Eating Behavior and Components of Body Composition and Metabolism in Adult Workers With Abdominal Obesity
Brief Title: Nutritional Counseling to Change Eating Behavior, Metabolism and Anthropometry in Adults With Abdominal Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Yolanda Fabiola Márquez Sandoval, Principal Investigator, University of Guadalajara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Universidad de Guadalajara
Record Dates: First submitted 2018-09-03; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Obesity, Abdominal
Keywords: obesity; nutritional counseling; weight loss; eating behaviors; abdominal obesity
MeSH Terms: conditions — Obesity, Abdominal; Obesity; Weight Loss; Feeding Behavior | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nutritional counseling (Experimental): Arm with intervention
  Interventions: Other: Nutritional counseling

INTERVENTIONS:
Other: Nutritional counseling — Intervention based on nutritional counseling under Cognitive Behavioral Theory and the used of strategies like self-monitoring, goals, cognitive restructuring and social support.

SUMMARY:
This study evaluates the impact of changes in eating behavior through nutritional counseling, after nine months of intervention, on body composition and metabolism in adult workers with abdominal obesity

DETAILED DESCRIPTION:
This study is a nutritional intervention in voluntary workers with abdominal obesity (waist circumference ≥102cm and ≥88cm). The intervention is divided into two phases: the intensive one has a duration of 6 months and consisted in a 4 face-to-face sessions with 9 online or telephone contacts based on the use of nutritional counseling [Academy of Nutrition and Dietetics, 2013] and the second phase: consisted in a 3 months' follow-up with 2 telephone contacts and a final visit face-to-face. The investigators used the Cognitive Behavior Therapy process as a theoretical framework, and also used the intervention comprised sessions designed to promote motivation, social support, self-regulation to promote the eating behavior change process. The participants were measured weight loss, waist circumference, and the lipid profile change, pre-intervention, and after six and nice months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* With abdominal obesity: men with waist circumference (CC) ≥102 cm and women with CC ≥88 cm.
* Literacy.
* Sign the informed consent

Exclusion Criteria:

* Participants with severe alterations of their renal function, hepatic, thyroid and circulatory system (self-reported or found in their laborarotorio analysis)
* Participants with any serious illness, hospitalization in the 6 months prior to the start of the study.
* In nutritional treatment for weight loss in the last three months.
* In psychological and / or psychiatric treatment.
* Depression or anxiety.
* History of bariatric surgery.
* Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2016-04-04 (Actual); Primary Completion 2017-08-12 (Actual); Study Completion 2018-01-17 (Actual)

PRIMARY OUTCOMES:
Change in eating behaviors | 6 and 9 months
  Increase consumption and frequency of healthy foods such as water, fruits and vegetables, healthy fats and fish. Decrease consumption and frequency of fatty foods, processed foods and sweet drinks. Evaluated by the validated tool Mini-ECCA.

SECONDARY OUTCOMES:
Anthropometric indicators | 6 and 9 months
  Decrease waist circumference
Decrease triglycerides | 6 and 9 months
  Decrease serum values of triglycerides

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda Fabiola Marquez Sandoval, PhD, Principal Investigator — University of Guadalajara

IPD SHARING:
Plan to Share IPD: No
The investigators will share only the global results to the participants, and company and university authorities for decision making.